CLINICAL TRIAL: NCT01901562
Title: Feasibility and Therapeutic Efficacy of Ductoscopic Papilloma Extraction in Patients With Pathologic Nipple Discharge
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not identify collaborator and secure additional funding following transfer of study to Montefiore Medical Center
Sponsor: Montefiore Medical Center (Other)
Collaborators: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAK3900
Record Dates: First submitted 2013-07-13; First posted 2013-07-17 (Estimated); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Breast Discharge Infected; Intraductal Papilloma of Breast
Keywords: ductoscopy; nipple discharge; breast; papilloma
MeSH Terms: conditions — Galactorrhea; Papilloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ductoscopic papillectomy (Experimental): Ductoscopic papillectomy to treat pathological nipple discharge
  Interventions: Device: Ductoscopic papillectomy

INTERVENTIONS:
Device: Ductoscopic papillectomy — Intraductal papilloma extraction through the nipple orifice by interventional ductoscopy

SUMMARY:
In this prospective clinical trial, patients who sign an approved informed consent for ductoscopy to assess etiology of Pathologic nipple discharge (PND) will be enrolled in the study. Consented patients who have been diagnosed with a solitary papilloma within the discharging duct will be recruited to have interventional ductoscopy.

Patients who are identified ductoscopically with a solitary non-sessile papilloma will undergo an attempted ductoscopic papillectomy (DP). Patients with ductoscopic findings other than single non-sessile papilloma will undergo standard ductoscopically guided microductectomy. The investigators will investigate whether the ductoscopic basket can be used as a safe endoscopic extraction instrument without adverse events. Histopathological evaluation will be performed to confirm the ductoscopic diagnosis and to determine the existence of any malignant tissue.

DETAILED DESCRIPTION:
Nipple discharge is the third most common breast related symptom for which women seek medical care, accounting for 37% of all breast complaints. Pathologic nipple discharge (PND) is defined as spontaneous or easily expressible single duct nipple discharge, which contributes to 5% of referrals to breast surgeons. Patients with PND represent a diagnostic and therapeutic challenge for the surgical clinician. The most frequent causes of PND in these cases are intraductal papilloma (IP) in 36% to 66%, ductal carcinoma in situ (DCIS) in 3% to 20% and other benign causes in up to 23%. The evaluation of women with PND usually involves radiological(mammography, ultrasound, ducto (galacto)graphy and cytological (nipple smear, ductal lavage) examinations; however, each of these procedures has found to have low sensitivity and specificity. A ductoscope is an instrument which allows visualization of abnormalities and polypoid lesions within the ductal system with access via the nipple orifice to aid in evaluation of PND. Moreover, it is currently being used to improve localization of lesions in patients with PND. Ductoscopically guided excision is an improvement over standard surgical approaches with terminal duct excision which removes a large volume of tissue with potential cosmetic deformity and for young women may make breast feeding not possible. Ductoscopy also allows retrieval of intraductal cells for diagnostic purposes using brush cytology.

ELIGIBILITY:
Inclusion Criteria:

* Be female
* Have pathologic (unilateral/uniductal) nipple discharge
* Been diagnosed with single papilloma
* Be over 18 years of age
* Sign the informed consent form

Exclusion Criteria:

* Have bilateral nipple discharge
* Personal history of breast cancer, ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS)
* Have BRCA 1 or 2 mutation
* Be currently pregnant or pregnant within the last 12 months
* Be currently lactating or lactated within the last 12 months
* Have received chemotherapy in the last 12 months
* Have had a Breast Imaging-Reporting and Data System (BIRADS) 3, 4, 5 or 6 mammograms within the last year
* Have diagnosed with multiple or sessile papilloma by ultrasound, mammography and/or ductoscopy.
* Have suspicious of malignancy in ultrasound
* Have an abnormal ﬁnding on the pre-operative nipple smear
* Have Gail Score >1.67
* Have had any subareolar or other surgery
* Have active infections or inﬂammation in a breast to be studied
* Have a known allergy to lidocaine
* Have abnormal liver function test
* Have medications know to be associated with breast discharge.
* Be unable to attend postoperative visits and imaging work-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09-27 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Feldman, MD, Principal Investigator — Montefiore Medical Center
Locations (2):
- United States (2):
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ductoscopic Papillectomy
Started | 9
Completed | 0
Not Completed | 9
Not completed — Protocol Violation | 5
Not completed — Excluded intraoperatively | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ductoscopic Papillectomy
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Complete Ductoscopic Retrievals
Description: Technical success will be determined by complete (total ductoscopic retrieval of a papilloma) ductoscopic retrieval of lesions over 90% of enrolled patients diagnosed with solitary papilloma.
Time Frame: 6 months
Population: Data related to the number of complete ductoscopic retrievals was not collected and analyzed.
Arm/Group | Ductoscopic Papillectomy
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Patients With Cessation of Nipple Discharge
Description: Therapeutic success will be determined by cessation after ductoscopic papillectomy (DP) in over 95% of enrolled patients with pathologic nipple discharge (PND) with a single papilloma.
Time Frame: Up to 2 weeks from the procedure
Population: Data related to the number of participants with cessation of nipple discharge after ductoscopic papillectomy was not collected and analyzed.
Arm/Group | Ductoscopic Papillectomy
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With Clinical Recurrence of Nipple Discharge
Description: Patients will be monitored for recurrence of nipple discharge at 6 month intervals for 2 years.
Time Frame: Up to 2 years
Population: Data related to the recurrence of nipple discharge was not collected and analyzed.
Arm/Group | Ductoscopic Papillectomy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months post treatment
Description: Five participants were excluded for not meeting protocol inclusion/exclusion criteria (i.e., screen failed) immediately following enrollment and did not participate in the study procedure.
  Four participants proceeded with the procedure. All four participants did not complete the study as the surgeon was unable to cannulate the ductal system or the patient was found to not have a solitary papilloma.
Arm/Group | Ductoscopic Papillectomy
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes